CLINICAL TRIAL: NCT03906591
Title: Evaluation Of Crestal Bone Level After Alveolar Bone Augmentation of Atrophied Posterior Mandibular Region Using Allogenic Bone Rings Vs. Autogenous Bone Rings With Simultaneous Dental Implant Placement (A Randomized Controlled Clinical Trial)
Brief Title: Crestal Bone Level After Allogenic Bone Ring With Simultaneous Dental Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa El-Deen Ragab Mahmoud, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: allogenic bone ring
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Allogenic Bone Ring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- allogenic bone ring (Experimental)
  Interventions: Procedure: allogenic bone ring
- autogenous bone ring (Active Comparator)
  Interventions: Procedure: autogenous bone ring

INTERVENTIONS:
Procedure: allogenic bone ring — allogenic bone ring with simultaneous dental implant placement
  Arms: allogenic bone ring
Procedure: autogenous bone ring — autogenous bone ring with simultaneous dental implant placement
  Arms: autogenous bone ring

SUMMARY:
This trial is aiming to answer a question whether in Patients with severely atrophied, distal mandibular regions, the use of allogenic bone rings with simultaneous dental implants, compared to autogenous bone rings, give successful clinical and radiographic outcomes without donor site morbidity

ELIGIBILITY:
Inclusion Criteria:

1. Medically free form any systemic diseases that contraindicate the surgical procedures or affect predictable outcomes and non-smoker subjects.
2. Atrophic mandibular distal region requiring vertical augmentation.
3. Good oral hygiene and healthy keratinized mucosa.

Exclusion Criteria:

1. Presence of acute dentoalveolar infection or any pathologic lesions.
2. Totally edentulous patients and patients requiring massive reconstruction and augmentation procedures.
3. Patients with history of previously failed augmentation procedures, or failed implant placement at the intended augmentation region.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
change in crestal bone height | at 6 months
  cone beam computed tomography will be used to measure bone height in millimeters

SECONDARY OUTCOMES:
graft failure | after 1 week, 6 months and after 9 months
  signs of graft failure will be evaluated by clinical examination
implant loss | after 1 week, 6 months and after 9 months
  signs of implant loss will be evaluated by clinical examination